CLINICAL TRIAL: NCT00402415
Title: A Phase I Trial of the Combination of Sirolimus and SU11248 (Sutent(R)) in Patients With Advanced Solid Tumors That Are Non-Curable With Standard Therapy
Brief Title: Study of Combination of Sirolimus and Sutent in Patients With Advanced Solid Tumors Non-Curable With Standard Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0510000723
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Tumors
Keywords: metastatic; malignancy; advanced solid tumors; unresectable; Solid Tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Sunitinib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sunitinib malate; Drug: Rapamycin

INTERVENTIONS:
Drug: Sunitinib malate — C1: 50 mg po days 1-15, 2 weeks off C2: 50 mg po x 4 weeks, 2 weeks off
  Other Names: SU11248; SUTENT®
Drug: Rapamycin — Dose escalation until MTD as follows:
  C1: not given C2: 4 mg weekly, 8 mg weekly, 12 mg weekly, 20 mg weekly
  Other Names: Sirolimus; Rapamune

SUMMARY:
There are two drugs involved in this study. Sunitinib (Sutent(R)) is approved by the Food and Drug Administration (FDA) for the treatment of advanced renal cell (kidney) cancer and gastrointestinal stromal tumors. Sunitinib is thought to work by blocking the growth of blood vessels into tumors; reducing the blood supply to tumors can slow their growth and sometimes causes the tumors to shrink. Sirolimus has been approved by the FDA to prevent the body from rejecting organ transplants. Sirolimus is being tested for its effects against cancer because it can slow the growth of some tumors in animal models. Sirolimus is thought to slow cancer growth in these animal models both by direct effects on the tumor cells, and also by blocking production of growth factors that stimulate production of blood vessels. We hope that the combined use of these two drugs will have better anti-cancer effects than either agent alone. This study is designed to find out if different doses of Sirolimus combined with a standard dose of Sutent are safe and well tolerated. Additionally, it is hoped to gain knowledge about the way that Sutent(R) in combination with sirolimus affects the blood vessels produced by cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. Patients with previously untreated metastatic renal cell carcinoma are eligible.
* Patients must have measurable disease by RECIST criteria.
* Patients must have at least 1 lesion located in the neck, lung, solid organ (including liver) or soft tissue in abdomen or pelvis, or soft tissue in lower extremities that is 3 cm and ideally <7 cm in the transaxial plane. Larger lesions may be considered if they meet all other criteria. Index lesions must be well demarcated.
* ECOG performance status of 0-1.
* Must be ≥18 years of age.
* Expected survival of at least 3 months.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Nursing patients are excluded. Sexually active men must also use acceptable contraceptive methods. Pregnant and nursing patients are excluded because the effects of the combination of SU11248 (Sutent®) and sirolimus on a fetus or nursing child are unknown.
* Must be able and willing to give written informed consent.
* Patients must have the following clinical laboratory values: ANC count ≥1500/mm3; Platelets ≥100,000/mm3; Serum creatinine ≤2x upper limit of normal. If serum creatinine is above the upper limit of normal (but less than 2x normal), patients must have a measured 24 hour urine creatinine clearance ≥ 50 ml/min to be eligible; Total bilirubin < 1.5x upper limit of normal; Serum calcium < 12.0 mg/dl; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3x the upper limit of normal; Prothrombin Time (PT), activated partial thromboplastin time (aPTT) and INR in the normal range;. Hemoglobin ≥9 gm/dl (may be corrected by transfusion).
* Normal cardiac ejection fraction

Exclusion Criteria:

* Diagnosis or history of central nervous system (CNS) disease (i.e. primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis).
* Any active uncontrolled bleeding and any patient with a bleeding diathesis (for example, active peptic ulcer disease). Any grade 3 hemorrhage within 4 weeks prior to starting treatment.
* Any ongoing coagulopathies or receiving anticoagulants.
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* QTc interval > 500 msec on baseline EKG.
* Cardiac ejection fraction below institutional lower limit of normal.
* Measured 24-hour urine creatinine clearance < 50 ml/min.
* Active infection of any kind.
* Unwilling or unable to follow protocol requirements or to give informed consent.
* Dyspnea at rest or with minimal exertion.
* No treatment with cytotoxic or biologic agents within the 4 weeks prior to beginning treatment on this study (6 weeks for mitomycin or nitrosoureas). At least 4 weeks must have elapsed from any prior surgery, radiation, hormonal or other drug therapy for their cancer. Patients must have fully recovered from the acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤ grade 1 are eligible.
* Any of the following within 6 months prior to first dose of treatment: myocardial infarction, symptomatic coronary artery disease (severe or unstable angina), artery bypass graft, uncontrolled arrhythmias, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolus.
* Known HIV infection. Patients with HIV infection are excluded because there may be unknown or dangerous drug interactions between sirolimus/SU11248 (Sutent®) and the anti-retroviral agents used to treat HIV infections.
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication.
* Diagnosis of second malignancy (except malignancies treated with no evidence of recurrence for at least 5 years, and curatively treated basal cell or squamous cell carcinomas of the skin, or in situ cervical cancer, or any stage I malignancy > 2 years from treatment).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Patients taking concurrent medications of any kind which are strong inducers or inhibitors of CYP3A4. Patients receiving any of the following will be excluded: ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's Wort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of sirolimus when combined with a standard dose and schedule of Sutent(R) | upon completion of dose escalation

SECONDARY OUTCOMES:
To obtain preliminary experience with dynamic MR imaging of tumor blood flow using the combination of Sutent(R) and sirolimus | upon completion of study
To provide preliminary data on dose effects of the combination on serum levels of VEGF and circulating endothelial cells | upon completion of study
To obtain preliminary information on the efficacy of Sutent(R)in combination with sirolimus in treating malignancies using RECIST criteria | upon completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut, United States